CLINICAL TRIAL: NCT06784349
Title: A Phase 1, Randomized, Double-Blind, Placebo-Controlled Study to Evaluate the Safety, Tolerability, Pharmacokinetics, and Pharmacodynamics of ALN-APOC3 in Adult Participants With Dyslipidemia
Brief Title: ALN-APOC3 in Adult Participants With Dyslipidemia
Status: Active, not recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Regeneron Pharmaceuticals (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Sequential | Masking: Quadruple | Purpose: Treatment
Other Study IDs: ALN-APOC3-hLP-2447
Record Dates: First submitted 2024-12-03; First posted 2025-01-20 (Actual); Last update posted 2025-12-29 (Actual); Status verified 2025-12

CONDITIONS: Dyslipidemia
Keywords: Lipids; Triglycerides; Cholesterol
MeSH Terms: conditions — Dyslipidemias

STUDY DESIGN:
Intervention Model Description: Part A: Sequential Part B: Parallel
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (5):
- ALN-APOC3 Ascending Cohorts (Experimental): Part A: Ascending Cohorts Randomized as described in the protocol May include optional cohorts
  Interventions: Drug: ALN-APOC3; Drug: Matching Placebo
- Placebo (Placebo Comparator): Part A and Part B:
  Randomized as described in the protocol
  Interventions: Drug: Matching Placebo
- ALN-APOC3 low-dose (Experimental): Part B: Parallel Arm Randomized as described in the protocol
  Interventions: Drug: ALN-APOC3
- ALN-APOC3 medium-dose (Experimental): Part B: Parallel Arm Randomized as described in the protocol
  Interventions: Drug: ALN-APOC3
- ALN-APOC3 high-dose (Experimental): Part B: Parallel Arm Randomized as described in the protocol
  Interventions: Drug: ALN-APOC3

INTERVENTIONS:
Drug: ALN-APOC3 — Administered as per the protocol
  Arms: ALN-APOC3 Ascending Cohorts; ALN-APOC3 high-dose; ALN-APOC3 low-dose; ALN-APOC3 medium-dose
Drug: Matching Placebo — Administered as per the protocol
  Arms: ALN-APOC3 Ascending Cohorts; Placebo

SUMMARY:
This study is researching an experimental drug called ALN-APOC3 (called "study drug"). The study is focused on participants who have dyslipidemia (abnormal amounts of fats in the blood, including triglycerides and cholesterol), but who are otherwise healthy.

The aim of the study is to see how safe and effective the study drug is.

The study is looking at several other research questions, including:

* What side effects may happen from taking the study drug
* How much study drug is in the blood at different times
* How the study drug changes lipid levels in the blood

ELIGIBILITY:
Key Inclusion Criteria:

1. Judged by the investigator to be in good health based on medical history, physical examination, vital signs, Electrocardiograms (ECG's) and laboratory safety testing, as defined in the protocol
2. Participants can enter the study under one of the following options, as defined in the protocol:

   1. Currently not taking statin and have not been on statin therapy for the 3 months prior to screening, or
   2. On a stable dose of statin, taken continuously for 3 months
3. Fasting triglycerides concentrations ≥100 and <500 mg/dL (1.13 to 5.65 mmol/L) during screening visit, as defined in the protocol
4. Fasting LDL-C ≥70 (1.81 mmol/L) if on stable statin therapy OR if not on statin treatment, as defined in the protocol

Key Exclusion Criteria:

1. History of clinically significant cardiovascular (other than dyslipidemia), respiratory, hepatic, renal, gastrointestinal, endocrine, hematological, psychiatric, or neurological disease, or any other concern, as assessed by the investigator that may confound the results of the study or poses an additional risk to the participant by study participation
2. Was hospitalized (ie, >24 hours) for any reason within 30 days of the screening visit
3. Is positive for Human Immunodeficiency Virus (HIV) or Hepatitis B surface Antigen (HBsAg) at the screening visit, as defined in the protocol
4. Is positive for hepatitis C antibody and positive for qualitative Hepatitis C Virus (HCV) Ribonucleic Acid (RNA) test at the screening visit
5. Any malignancy, except for non-melanoma skin cancer or cervical/anus in-situ, that have been resected with no evidence of metastatic disease for 3 years prior to the screening visit

NOTE: Other protocol defined inclusion/exclusion criteria apply

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 32 (Actual)
Dates: Start 2025-01-27 (Actual); Primary Completion 2026-02-25 (Estimated); Study Completion 2026-02-25 (Estimated)

PRIMARY OUTCOMES:
Incidence of Treatment Emergent Adverse Events (TEAEs) | Through Week 44
Severity of TEAEs | Through Week 44
Percent changes in fasting concentrations of High-Density Lipoprotein Cholesterol (HDL-C) | Baseline to week 24
  Part B Only

SECONDARY OUTCOMES:
Concentration of combined ALN-APOC3 and metabolites in plasma | Through Week 44
Urinary excretion of combined ALN-APOC3 and metabolites | Through 24 Hours, After Treatment
  Part A Only
Percent change in fasting concentrations of APOC3 | Baseline to Week 12
Absolute change in fasting concentrations of APOC3 | Baseline to Week 12
Percent change in fasting concentrations of APOC3 | Baseline to Week 24
  Part B Only
Absolute change in fasting concentrations of APOC3 | Baseline to Week 24
  Part B Only
Percent change in fasting concentrations of HDL-C | Baseline to Week 12
Absolute change in fasting concentrations of HDL-C | Baseline to Week 12
Absolute change in fasting concentrations of HDL-C | Baseline to Week 24
  Part B Only
Percent change in fasting concentrations of Low-Density Lipoprotein Cholesterol (LDL-C) | Baseline to Week 12
Absolute change in fasting concentrations of LDL-C | Baseline to Week 12
Percent change in fasting concentrations of LDL-C | Baseline to Week 24
  Part B Only
Absolute change in fasting concentrations of LDL-C | Baseline to Week 24
  Part B Only
Percent change in fasting concentrations of Triglycerides (TG) | Baseline to Week 12
Absolute change in fasting concentrations of TG | Baseline to Week 12
Percent change in fasting concentrations of TG | Baseline to Week 24
  Part B Only
Absolute change in fasting concentrations of TG | Baseline to Week 24
  Part B Only
Percent change in fasting concentrations of non-HDL-C | Baseline to Week 12
Absolute change in fasting concentrations of non-HDL-C | Baseline to Week 12
Percent change in fasting concentrations of non-HDL-C | Baseline to Week 24
  Part B Only
Absolute change in fasting concentrations of non-HDL-C | Baseline to Week 24
  Part B Only
Percent change in fasting concentrations of Apolipoprotein-B (APOB) | Baseline to Week 12
Absolute change in fasting concentrations of APOB | Baseline to Week 12
Percent change in fasting concentrations of APOB | Baseline to Week 24
  Part B Only
Absolute change in fasting concentrations of APOB | Baseline to Week 24
  Part B Only

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Trial Management, Study Director — Regeneron Pharmaceuticals
Locations (1):
- Arensia Exploratory Medicine at the Republican Clinical Hospital, Chisinau, Moldova

IPD SHARING:
Plan to Share IPD: Yes
All Individual Patient Data (IPD) that underlie publicly available results will be considered for sharing.
Supporting Information: Study Protocol, SAP, ICF, CSR, Analytic Code
Time Frame: When Regeneron has:
  * received marketing authorization from major health authorities (e.g., FDA, European Medicines Agency (EMA), Pharmaceuticals and Medical Devices Agency (PMDA), etc.) for the product and indication or has globally discontinued development of the product for all indications on or after April 2020 and has no plans for future development
  * made the study results publicly available (e.g., scientific publication, scientific conference, clinical trial registry)
  * the legal authority to share the data, and
  * ensured the ability to protect participant privacy
Access Criteria: Qualified researchers can submit a proposal for access to individual patient or aggregate level data from a Regeneron-sponsored clinical trial through Vivli. Regeneron's Independent Research Request Evaluation Criteria can be found at: https://www.regeneron.com/sites/default/files/Regeneron-External-Data-Sharing-Policy-and-Independent-Research-Request-Evaluation-Criteria.pdf
URL: https://vivli.org/